CLINICAL TRIAL: NCT01003587
Title: Improving Use of Evidence in Policy: District Evaluation Study on Health
Brief Title: Promoting Evidence-Based Decision-Making in India: District Evaluation Study on Health
Acronym: DESH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian International Development Agency (Other Government); Lombard Insurance Global Poverty Action Lab (Unknown); St. John's Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SMH 09-049
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Infectious Disease; Cardiovascular Disease
Keywords: India; evidence-based policy; knowledge translation; disease control priorities; decision-makers; health spending; health services delivery; maternal and child health; policy making; delivery of health care
MeSH Terms: conditions — Communicable Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- District health information package (Experimental)
  Interventions: Behavioral: District health information package
- No Intervention (No Intervention)

INTERVENTIONS:
Behavioral: District health information package — The intervention package consists of:
  * A report on disease burden, disease control priorities and health system performance in India
  * Condensed fact sheet based on the report
  * District health report cards (DRCs) comparing performance on key health indicators with other districts, information on causes of death in each district, and actionable messages to reduce deaths in the district
  * Customized speech for district level officials detailing key actions to reduce deaths
  * Reminder materials including poster version of the DRCs and video on key points and actionable messages
  Arms: District health information package

SUMMARY:
The purpose of this study is to assess the impact of disseminating information on comparative performance, along with actionable messages on how to improve health outcomes, to district-level decision-makers in India using a randomized, controlled design. This information should improve prioritization of health services by district health officers, budget allocation for health, and implementation of priority health services at the district level.

DETAILED DESCRIPTION:
Use of evidence in policy is uneven, leading to frequent waste of resources. However, the best way to promote evidence uptake in policy formulation and implementation is unclear. Information on disease control priorities based on India's disease burden and health system capacity has been produced to help focus government efforts during a period of increased spending and decentralization.

This study tests the impact of sending information on comparative performance (using district report cards) and actionable messages (on how to reduce disease burden) to district-level decision-makers on uptake of disease control priority recommendations in India. Using a cluster-randomized design, districts will be randomized to receive either the mailed information package or no intervention. The sample includes all 594 Indian districts in existence in 2001. The intervention will target key district level decision-makers: parliamentarians (Members of Parliament, Members of Legislative Assembly), bureaucrats (District Collectors), technocrats (District Health Officers), and local government officials (Zilla Parishad CEOs).

Study outcome data will be collected using sequential national surveys of health service availability and utilization, including relevant rounds of the District Level Health and Facility Surveys and the Annual Health Surveys. This study tests an inexpensive, pragmatic strategy on a large scale and will provide information on effective methods of knowledge translation to policy-makers.

ELIGIBILITY:
Inclusion Criteria (Districts):

* All districts in India in existence in 2001

Exclusion Criteria (Districts):

* All districts in India created after 2001

Inclusion Criteria (District Officials):

* Members of Parliament (MPs) who sit in the Lok Sabha (Lower House of Parliament) and represent constituencies that are contained within or overlap study districts
* Members of Legislative Assembly (MLAs) who represent constituencies that are contained within study districts
* District Collectors (DCs) who administrate study districts
* Zilla Parishad Chief Executive Officers (ZPCEOs) who administrate study districts
* District Health Officers (DHOs) who work in study districts

Exclusion Criteria (District Officials):

* MPs who sit in the Rajya Sabha (Upper House of Parliament), Lok Sabha MPs who represent constituencies not contained within or overlapping study districts, Lok Sabha MPs who represent constituencies that overlap both experimental and control study districts
* MLAs who represent constituencies not contained within study districts
* DCs who administrate non-study districts
* ZPCEOs who administrate non-study districts
* DHOs who work in non-study districts

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2009-07; Primary Completion 2016-03 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Percentage children 12-23 months vaccinated against measles | Five years
Percentage children <3 yrs with diarrhea in past 2 weeks given oral rehydration solution | Five years
Percentage facility-based births for the last child since 2007 | Five years

SECONDARY OUTCOMES:
Percentage last child >3 yrs breast fed within 1 hr of birth | Five years
Percentage women given advice on breastfeeding and newborn thermal care during antenatal care | Five years
Percentage subcenters with oral rehydration solution available on day of survey and no stockouts for more than 10 days in last month | Five years
Percentage community health centres with at least 1 surgeon or ob/gyn | Five years
Percentage public health centres with reagents, light microscope and lab technician for malaria blood smear | Five years

OTHER OUTCOMES:
Differences in any of primary and secondary outcomes between Empowered Action Group and Assam (EAGA) states and non-EAGA states | Five years
Differences in any of primary and secondary outcomes between measles-focus states and non-measles-focus states | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Onil Bhattacharyya, MD, PhD, Principal Investigator — Unity Health Toronto; Prabhat Jha, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (2):
- Centre for Global Health Research, St. Michael's Hospital, Toronto, Ontario, Canada
- St. John's Research Institute, Bangalore, Karnataka, India

REFERENCES:
- See also: Centre for Global Health Research — http://www.cghr.org
- See also: St. John's Research Institute — http://www.sjri.res.in/